CLINICAL TRIAL: NCT04168697
Title: The Effect of Behavioral Intervention on the Cannabinoid Receptor System in Patients With Bipolar Affective Disorder
Brief Title: Effect of Behavioral Intervention on Cannabinoid Receptors in BAD
Acronym: WHM_BAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Otto Muzik, Professor of Pediatrics, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19061167
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Bipolar Affective Disorder, Currently in Remission; Bipolar Disorder I; Bipolar Disorder II
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Patient group vs a control group
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Experimental): Control subjects undergoing an 8-week behavioral modification technique consisting of a combination of breathing exercises, cold exposure and meditation
  Interventions: Behavioral: Wim Hof method
- BAD (Experimental): Patients with bipolar affective disorder (BAD) undergoing an 8-week behavioral modification technique consisting of a combination of breathing exercises, cold exposure and meditation
  Interventions: Behavioral: Wim Hof method

INTERVENTIONS:
Behavioral: Wim Hof method — 8-week behavioral modification intervention instructing the participants in a combination of breathing exercises, cold exposure and meditation

SUMMARY:
The objective of this study is to determine whether the practice of a non-drug related intervention technique (behavioral modification technique consisting of a combination of breathing exercises, cold exposure and meditation) has an effect on long-term cannabinoid receptor function in a control group as well as in a group of patients suffering from bipolar affective disorder (BAD). Specifically, the objective of this study is to test whether the applied behavioral modification technique is able to alter cannabinoid receptor density in brain areas that modulate mood and motivational drive (such as vmPFC, PAG, VTA, amygdala and OFC). The investigators believe that these studies will form the impetus for a better understanding and deployment of non-drug related treatment methods in patients with various depressive symptoms. In particular, it appears that the proposed behavioral modification technique might be a powerful, currently under-appreciated, method to positively modulate the brain's own cannabinoid system.

DETAILED DESCRIPTION:
Bipolar affective disorder (BAD) is often poorly controlled by prescribed drugs. Clinical observations suggest that the endocannabinoid system is dysfunctional in BAD and fails to control the level of cortical excitation and inhibition in the brain. Thus, excessively high endocannabinoid tone (mania) or excessively low endocannabinoid tone (depression) may manifest itself in BAD patients. Interestingly, cannabis use is common in patients with this disorder and anecdotal reports suggest that some patients take it to alleviate symptoms of both mania and depression. The investigators have recently studied brain activations during a cold stress paradigm in a 57 year old Dutch national (Wim Hof), the so-called "Iceman", who has the ability to withstand frequent prolonged periods of extreme cold exposure using a self-developed technique that includes a combination of breathing exercises, cold exposure and meditation (referred to as the WH technique). The WH technique allows the "Iceman" to regulate his own autonomic nervous system in the presence of severe cold and to perform remarkable acts of survival under extreme thermal conditions. Moreover, it has been shown that the WH technique can be successfully taught to novice users. Preliminary studies performed by the investigators have examined CNS mechanisms associated with the practice of the WH technique and the obtained findings unequivocally demonstrated activation of autonomic brainstem areas that are implicated in stress-induced analgesia as well as cognitive cortical areas that are associated with self-reflection (such as the anterior insula). In particular, a strong activation of the periaqueductal gray (PAG) was determined, which is implicated in the release of endogenous opiates/cannabinoids that mediate decreased sensitivity to cold exposure and (via connections to higher-order cortical areas) promote a feeling of euphoria and well-being. This finding suggests that the WH technique might allow practitioners to assert increased level of control over key components of the affective system and as a result might be a viable, non-drug related approach for patients with pathological mood swings. The investigators believe that this method might be particularly effective in patients suffering from BAD, as the practice of the WH technique can be implemented during both remission and at the onset of highly motivational manic episodes, which will then help to limit the effects of negative mood swings during depressive (and manic) episodes. The investigators will study the effects of the WH technique on cannabinoid receptor density using the cannabinoid PET tracer (F18-FMPEP-d2) by determining regional changes in cannabinoid receptor density in various brain regions prior and post behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

* BAD type I or II, in clinical remission of acute mood episode at least 3 months prior to study
* Having experienced an acute affective episode in the past 3 years
* Having suffered at least two lifetime depressive episodes
* Monotherapy or combination with a mood stabilizer (lithium, valproate, carbamazepine or lamotrigine) at optimal doses, quetiapine monotherapy or in combination with the aforementioned stabilizers, any oral atypical antipsychotic in combination with an antidepressant
* Hamilton Depression Rating Scale (HDRS) score (>8 and <19) and Young Mania Rating Scale (YMRS) score <10
* Being able to understand and agree with requirements of study protocol

Exclusion Criteria:

* (i) Any acute mood episode in the 12 weeks before the start of the trial
* Any current DSM-IV diagnosis different from BAD (including substance or alcohol use disorder at the time of study entry, except if it is under complete remission. Not applicable to nicotine or caffeine)
* Risk of suicide or self/hetero aggressiveness
* Pregnancy
* Severe and unstable medical disease
* Mental retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Cannabinoid PET imaging | 12 weeks
  Changes in cannabinoid receptor density measured using F18-FMPEP-d2 PET/CT imaging pre and post behavioral intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
At this to we plan to share only summary data that will be published in peer-reviewed journals.